CLINICAL TRIAL: NCT04084288
Title: Intraoperative Acupuncture for Low-Dose Opioid Total Knee Replacement: An Observational Prospective Cohort Study
Brief Title: Acupuncture for Low-Dose Opioid for TKA Replacement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-1193
Record Dates: First submitted 2019-09-09; First posted 2019-09-10 (Actual); Results first posted 2022-05-05 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-09

CONDITIONS: Knee Osteoarthritis; Pain, Postoperative; Acupuncture
Keywords: Acupuncture, Total Knee Replacement
MeSH Terms: conditions — Osteoarthritis, Knee; Pain, Postoperative | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Postoperative Acupuncture (Experimental): Neuraxial anesthesia (spinal or combined spinal epidural (CSE) with up to 4cc mepivacaine 1.5%) and 2 blocks for postoperative pain (IPACK and adductor canal peripheral nerve blocks). Sedation will be provided. Tranexemic acid (TXA) will be dosed per surgeon request.
  A certified medical acupuncturist will perform ipsilateral Auricular Trauma Protocol (ATP) acupuncture at eight ear points (Hypothalamus, Amygdala, Hippocampus, Prefrontal Cortex, Point Zero, Shen Men, Insula, Vagus) with 30Hz electrostimulation at two of those points (Shen Men and Hypothalamus). Acupuncture needles will be left in place and stimulated for 60 min and then removed. If an epidural is placed, it may be redosed with lidocaine as needed (up to 100mg total) and will be removed prior to transfer to the recovery room.
  A periarticular injection (PAI) will be placed by the surgeon during the surgery (timing at the discretion of the surgeon)
  Interventions: Other: Acupuncture; Device: Peripheral Nerve Stimulator

INTERVENTIONS:
Other: Acupuncture — Ipsilateral Auricular Trauma Protocol (ATP) acupuncture at eight ear points (Hypothalamus, Amygdala, Hippocampus, Prefrontal Cortex, Point Zero, Shen Men, Insula, Vagus) with 30Hz electrostimulation at two of those points (Shen Men and Hypothalamus). Acupuncture needles will be left in place and stimulated for 60 min and then removed
Device: Peripheral Nerve Stimulator — Ipsilateral Auricular Trauma Protocol (ATP) acupuncture at eight ear points (Hypothalamus, Amygdala, Hippocampus, Prefrontal Cortex, Point Zero, Shen Men, Insula, Vagus) with 30Hz electrostimulation at two of those points (Shen Men and Hypothalamus).

SUMMARY:
The majority of patients undergoing total knee replacement(TKR) rely on opioids for postoperative analgesia. These medications have undesirable side effects and potential for abuse and addiction. The aim of this cohort study is to determine the incidence rate of patients who are able to maintain a low dose opioid regimen after TKR with the use of a multimodal approach that includes intraoperative auricular acupuncture protocol.

DETAILED DESCRIPTION:
This is a prospective cohort study to assess the feasibility of patients to undergo TKR while adhering to a low-dose opioid regimen by using a multimodal analgesic approach that includes intraoperativeauricular acupuncture. We hypothesize that it will be feasible to maintain a low-dose opioid regimen during TKR while followingthe intraoperative auricular acupuncture protocol, and that patients will be satisfied with their pain control with a low incidence of adverse events.

ELIGIBILITY:
Inclusion Criteria:

* ASA of 1 or 2
* Age 18-70
* Undergoing primary total knee replacement
* Desire to attempt a low opioid or opioid free pathway

Exclusion Criteria:

* NonEnglish speaking
* Patients with the inability to understand or follow study protocol
* Opioid use in the last 6 weeks or chronic pain patient
* Cannot receive neuraxial anesthesia and/or peripheral nerve block
* Patients with contraindications to intraop protocol (e.g., patient cannot take acetaminophen or ketorolac due to liver or kidney disease)
* Patients with implanted cardiac device such as a pacemaker or AICD
* Active ear infection
* Nonnative ear, previous scarring or surgical manipulation of ear
* Patients with gauges or other deforming ear piercing (small nondeforming ear piercings are ok) present in ears
* Allergy to nickel

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2019-08-21 (Actual); Primary Completion 2020-10-02 (Actual); Study Completion 2020-10-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Cheng, MD, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices)
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Beginning 3 months and ending 5 years following article publication.
Access Criteria: Researchers who provide a methodologically sound proposal. This will be done to achieve aims in the approved proposal. Proposals should be directed to chengs@hss.edu. To gain access, data requestors will need to sign a data access agreement. Data are available for 5 years at a third party website.

RESULTS

PARTICIPANT FLOW:
Groups:
- Postoperative Acupuncture: Neuraxial anesthesia (spinal or combined spinal epidural (CSE) with up to 4cc mepivacaine 1.5%) and 2 blocks for postoperative pain (IPACK and adductor canal peripheral nerve blocks). Sedation will be provided. Tranexemic acid (TXA) will be dosed per surgeon request.
  A certified medical acupuncturist will perform ipsilateral Auricular Trauma Protocol (ATP) acupuncture at eight ear points (Hypothalamus, Amygdala, Hippocampus, Prefrontal Cortex, Point Zero, Shen Men, Insula, Vagus) with 30Hz electrostimulation at two of those points (Shen Men and Hypothalamus). Acupuncture needles will be left in place and stimulated for 60 min and then removed. If an epidural is placed, it may be redosed with lidocaine as needed (up to 100mg total) and will be removed prior to transfer to the recovery room.
  A periarticular injection (PAI) will be placed by the surgeon during the surgery (timing at the discretion of the surgeon)
  Acupuncture: Ipsilateral Auricular Trauma Protocol (ATP) acupuncture at eight ear points (Hypothalamus, Amygdala, Hippocampus, Prefrontal Cortex, Point Zero, Shen Men, Insula, Vagus) with 30Hz electrostimulation at two of those points (Shen Men and Hypothalamus). Acupuncture needles will be left in place and stimulated for 60 min and then removed
Period: Overall Study
Arm/Group | Postoperative Acupuncture
Started | 41
Completed | 41
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Postoperative Acupuncture
Number analyzed (Participants) | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.9 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 39
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 34
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 41

OUTCOME MEASURES:

1. Primary Outcome: Low-dose Opioid Regimen Adherence
Description: The number of patients who maintain a low-dose opioid regimen (15 pills or less of 5mg oxycodone or 112.5 OME [oral morphine equivalents]) from postoperative day (POD) 0 to POD 30 throughout their Total Knee Replacement.
Time Frame: postoperative day 0 to postoperative day 30
Measure: Number; unit: participants
Arm/Group | Postoperative Acupuncture
Number analyzed (Participants) | 41
participants | 26

2. Secondary Outcome: Total Opioid Consumption
Description: Postoperative opioid consumption measured in oral morphine equivalents (OME) at various timepoints
Time Frame: post anesthesia care unit (PACU), postoperative day (POD) 1, POD7, POD14, POD30
Population: One patient lost to follow-up on POD1.
Measure: Mean (Standard Deviation); unit: oral morphine equivalents (OME)
Arm/Group | Postoperative Acupuncture
Number analyzed (Participants) | 41
oral morphine equivalents (OME)
  PACU | 14.9 (12.4)
  POD1: number analyzed (Participants) | 40
  POD1 | 11.9 (20)
  POD2: number analyzed (Participants) | 40
  POD2 | 7.3 (15.5)
  POD7: number analyzed (Participants) | 40
  POD7 | 13.5 (55.7)
  POD14: number analyzed (Participants) | 40
  POD14 | 108.3 (190.4)
  POD30: number analyzed (Participants) | 40
  POD30 | 0 (0)

3. Secondary Outcome: Numerical Rating Scale (NRS) Pain Scores at Rest and With Movement
Description: Numerical Rating Scale (NRS) pain scores at rest and with movement. NRS pain is measured from 0 to 10, with 0 being the no pain whatsoever and 10 being the worst pain imaginable.
Time Frame: post anesthesia care unit (PACU), postoperative day (POD) 1, POD7, POD14, POD30
Population: One patient lost to follow-up on POD1. Some patients were not available for administration of NRS at all time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Postoperative Acupuncture
Number analyzed (Participants) | 41
score on a scale
  Pre-Op: number analyzed (Participants) | 39
  Pre-Op | 5.1 (2.2)
  POD0: number analyzed (Participants) | 39
  POD0 | 4.2 (2.7)
  POD1: number analyzed (Participants) | 39
  POD1 | 3.7 (2)
  POD7: number analyzed (Participants) | 38
  POD7 | 3.7 (2.2)
  POD14: number analyzed (Participants) | 35
  POD14 | 3 (1.8)
  POD30: number analyzed (Participants) | 37
  POD30 | 2.4 (1.9)

4. Secondary Outcome: Duration of Neuraxial Anesthesia in Hours
Description: Duration of neuraxial anesthesia is defined as number of hours between anesthesia start time to anesthesia stop time.
Time Frame: postoperative day 1
Population: Duration of neuraxial anesthesia in hours
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Postoperative Acupuncture
Number analyzed (Participants) | 41
Hours | 2.6 (0.3)

5. Secondary Outcome: Deviation From Prescribed Oral Pain Regimen
Description: Tracking the number of patients that received different oral pain main medication, including the need for rescue medications by postoperative day 30
Time Frame: Postoperative day 30
Measure: Count of Participants; unit: Participants
Groups:
- Postoperative Acupuncture: Neuraxial anesthesia (spinal or combined spinal epidural (CSE) with up to 4cc mepivacaine 1.5%) and 2 blocks for postoperative pain (IPACK and adductor canal peripheral nerve blocks). Sedation will be provided. Tranexemic acid (TXA) will be dosed per surgeon request. A certified medical acupuncturist will perform ipsilateral Auricular Trauma Protocol (ATP) acupuncture at eight ear points (Hypothalamus, Amygdala, Hippocampus, Prefrontal Cortex, Point Zero, Shen Men, Insula, Vagus) with 30Hz electrostimulation at two of those points (Shen Men and Hypothalamus). Acupuncture needles will be left in place and stimulated for 60 min and then removed. A periarticular injection (PAI) will be placed by the surgeon during the surgery (timing at the discretion of the surgeon) Acupuncture: Ipsilateral Auricular Trauma Protocol (ATP) acupuncture at eight ear points (Hypothalamus, Amygdala, Hippocampus, Prefrontal Cortex, Point Zero, Shen Men, Insula, Vagus) with 30Hz electrostimulation at two of those points (Shen Men and Hypothalamus). Acupuncture needles will be left in place and stimulated for 60 min and then removed Peripheral Nerve Stimulator: Ipsilateral Auricular Trauma Protocol (ATP) acupuncture at eight ear points (Hypothalamus, Amygdala, Hippocampus, Prefrontal Cortex, Point Zero, Shen Men, Insula, Vagus) with 30Hz electrostimulation at two of those points (Shen Men and Hypothalamus).
Arm/Group | Postoperative Acupuncture
Number analyzed (Participants) | 41
Participants
  Lost to Follow up | 1
  Protocol Deviations | 0

6. Secondary Outcome: Number of Participants With Side Effects on POD1 and During the PACU Stay
Description: Incidence of nausea, vomiting, pruritus (itching), and constipation. These are reported by the patient in the PACU and on postoperative day 1
Time Frame: PACU, Postoperative day 1
Population: Patients who answer yes to side effects in the past 24hr for POD1
Measure: Number; unit: participants
Groups:
- Side Effects in the Past 24 hs POD 1: for POD 1, In the last 24 hours, have you had any nausea, vomiting, constipation, difficulty passing urine, concentrating, staying awake, lightheaded/dizzy, confused, general fatigue, itchiness, dry mouth, headache?
- Side Effects PACU: Incidence of nausea, vomiting, pruritus, constipation reported in the PACU by patient
Arm/Group | Side Effects in the Past 24 hs POD 1 | Side Effects PACU
Number analyzed (Participants) | 41 | 41
participants
  Nausea | 11 | 7
  Vomiting | 4 | 0
  Constipation | 3 | 0
  Difficulty passing urine | 2 | 3
  Concentrating | 2 | 1
  Drowsy/staying awake | 8 | 9
  Lightheaded or Dizzy | 8 | 9
  Confused | 2 | 0
  General fatigue/weaknesses | 7 | 6
  Itchiness | 4 | 0
  Dry mouth | 15 | 16
  Headache | 7 | 0

7. Secondary Outcome: Postoperative Range of Motion
Description: Postoperative range of motion measured at the 6 week surgeon office visit. This is being measured by either the physician or their PA and is a score that is achieved by adding extension and flexion together. It is measured in degrees. (example: flexion: 118 + extension:1 = score: 119)
Time Frame: 6 weeks postoperative (surgeon office visit)
Population: 6 weeks post-op follow up. Only 5 patients completed this secondary measure.
Measure: Mean (Standard Deviation); unit: degrees
Groups:
- Knee Range of Motion (ROM) at 6 Weeks: Range of motion at 6 weeks F/U for surgery
Arm/Group | Knee Range of Motion (ROM) at 6 Weeks
Number analyzed (Participants) | 5
degrees | 113.2 (20.5)

8. Secondary Outcome: Tourniquet Time
Description: Duration of time the tourniquet is inflated intraoperatively. Measured in minutes
Time Frame: Intraoperatively
Population: Length of time for tourniquet inflated during the intra-operative. 5 patients out of 41 did not have tourniquets.
Measure: Mean (Standard Deviation); unit: minutes
Groups:
- Tourniquet Intra-operative: Length of tourniquet time during intra-operative
Arm/Group | Tourniquet Intra-operative
Number analyzed (Participants) | 36
minutes | 60.5 (11.7)

ADVERSE EVENTS:
Time Frame: The duration of patient enrollment (1 year)
Arm/Group | Postoperative Acupuncture
All-Cause Mortality (participants affected / at risk) | 0/41
Serious Adverse Events (participants affected / at risk) | 0/41
Other Adverse Events (participants affected / at risk) | 0/41

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-24): https://cdn.clinicaltrials.gov/large-docs/88/NCT04084288/Prot_SAP_002.pdf